CLINICAL TRIAL: NCT02406573
Title: A Pilot Study to Assess Nominal Versus Controlled Stimuli on Dentinal Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015024
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Dentin Sensitivity
Keywords: Sensitivity
MeSH Terms: conditions — Dentin Sensitivity; Hypersensitivity

ARMS (1):
- Crest® Sensi-Stop™ Strips (Experimental): Professionally Applied
  Interventions: Device: Crest® Sensi-Stop™ Strips

INTERVENTIONS:
Device: Crest® Sensi-Stop™ Strips

SUMMARY:
This pilot study will evaluate the use of nominal stimuli to assess dentinal hypersensitivity response relative to a clinically-controlled stimulus.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age
* sign an informed consent form and be given a copy
* be in good general health as determined by the Investigator/designee
* agree to delay any elective dentistry, including dental prophylaxis, and to report any dentistry received during the course of the study
* agree to not participate in any other oral care study for the duration of this study
* agree to return for scheduled visits and follow all study procedures
* have dentinal hypersensitivity with at least one tooth with a Schiff sensitivity score of at least 1 in response to the examiner applied cold water challenge

Exclusion Criteria:

* severe periodontal disease, as characterized by purulent exudate, generalized mobility, and/or severe recession
* active treatment for periodontitis
* any diseases or conditions that might interfere with the subject safely completing the study
* inability to undergo study procedures
* fixed facial orthodontic appliances
* a history of kidney stones
* self-reported pregnancy or nursing
* known allergies to the following ingredients; aqua, glycerin, cellulose gum, dipotassium oxalate, carbomer, sodium hydroxide, sodium benzoate, and potassium sorbate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Gerlach, DDS, MPH, Principal Investigator — Procter and Gamble
Locations (1):
- Oral Health Science Center, Mason, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Crest® Sensi-Stop™ Strips: Professionally Applied
  Crest® Sensi-Stop™ Strips
Period: Overall Study
Arm/Group | Crest® Sensi-Stop™ Strips
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Crest® Sensi-Stop™ Strips
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (7.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian Oriental | 2
  Black | 3
  Caucasian | 24
  Asian Indian | 1
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline for Visual Analog Scale - Cold Water
Description: Visual Analog Scale (VAS) - subjects are asked to look at a VAS and designate the level of hypersensitivity they experienced as a result of the thermal and water challenges using a continuum scale of 0 = No tooth pain up to 100 = Worst tooth pain ever experienced.
Time Frame: Day 1
Population: Thirty (30) subjects received study product and completed the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crest® Sensi-Stop™ Strips
Number analyzed (Participants) | 30
Units on a scale | -22.93 (31.10)

2. Primary Outcome: Change From Baseline for Dentin Sensitivity Cold Water as Assessed by the Schiff Index
Description: The Schiff Sensitivity Scale was assessed for each test tooth via an evaporative air challenge. The examiner recorded the Schiff Index score corresponding to the response to the air challenge. The Schiff Index Sensitivity scale is scored as follows- 0: tooth/subject did not respond to stimulus, 1: tooth/subject responds to stimulus, but does not request discontinuation of stimulus, 2: tooth/subject responds to stimulus and requests discontinuation or moves form stimulus, 3: tooth/subject responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. The higher the Schiff score, the more sensitive the tooth. The mean change from Baseline was calculated for this measure.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crest® Sensi-Stop™ Strips
Number analyzed (Participants) | 30
Units on a scale | -0.17 (0.79)

3. Primary Outcome: Change From Baseline for 5 Face Emoticon Scale
Description: Scale to score their comfort/discomfort that ranges from -2 to +2 where a -2 is considered very comfortable and a +2 is considered very uncomfortable.
Time Frame: Day 2
Population: Thirty (30) subjects received study product and completed the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Crest® Sensi-Stop™ Strips
Number analyzed (Participants) | 30
Units on a scale | -1.07 (1.53)

ADVERSE EVENTS:
Arm/Group | Crest® Sensi-Stop™ Strips
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 7/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crest® Sensi-Stop™ Strips (N=30)
Gingivitis (Gastrointestinal disorders) | 4 (4)
Mucous Mem Dis (Gastrointestinal disorders) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes